CLINICAL TRIAL: NCT05069753
Title: Patient Reported Visual Function Outcome Following Bilateral Cataract Surgery
Brief Title: Patient Reported Visual Satisfaction Following Same Day or Delayed Bilateral Cataract Surgery
Acronym: CatquestCBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mads Assenholt Nielsen, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CatQuestCBS
Record Dates: First submitted 2021-09-14; First posted 2021-10-06 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Bilateral Cataract; Charles Bonnet Syndrome
MeSH Terms: conditions — Cataract; Charles Bonnet Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of two groups using a digital coin toss. Thus they will either undergo same day-surgery of both eyes or have the two surgical procedures separated by one week.
Masking Description: No masking: The patients will be informed of the type of procedure they will undergo.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate sequential bilateral cataract surgery (ISBCS) (Active Comparator)
  Interventions: Procedure: Immediate sequential bilateral cataract surgery (ISBCS)
- Delayed sequential bilateral cataract surgery (DSBCS) (Active Comparator)
  Interventions: Procedure: Delayed sequential bilateral cataract surgery (DSBCS)

INTERVENTIONS:
Procedure: Immediate sequential bilateral cataract surgery (ISBCS) — Surgery on both eyes will be performed on the same day as separate procedures: Once surgery on the first eye is completed, a new sterile procedure on the second eye will commence.
  Arms: Immediate sequential bilateral cataract surgery (ISBCS)
Procedure: Delayed sequential bilateral cataract surgery (DSBCS) — The group will undergo bilateral cataract surgery on two separate days with a time period of one week between the two procedures.
  Arms: Delayed sequential bilateral cataract surgery (DSBCS)

SUMMARY:
Cataract is currently the leading cause of visual impairment worldwide with age being the most common cause of lenticular opacification. As cataract surgery is the most commonly performed elective surgery worldwide, forecasts of an increasing number of elderly individuals make it clear that efficient and evidence based models for managing cataract in the future need to be implemented to manage the broadening gap between intervention and available resources.

Bilateral cataract is currently treated using same day separate surgical procedures (immediate sequential bilateral cataract surgery (ISBCS) or on separate days (delayed sequential bilateral cataract surgery (DSBCS). Whether one approach is more ideal than the other is an ongoing debate. There is, however, a clear advantage of same day surgery on resource management.

The primary purpose of this clinical study is to measure the patient reported satisfaction regarding vision in a group of 300 participants following either same day or delayed bilateral cataract surgery.

DETAILED DESCRIPTION:
In this study, patient reported satisfaction in regards to vision is measured using a questionnaire based on the validated Catquest-7SF questionnaire. This is a 7-item self-report scale with both general questions related to difficulties in performing daily activities and satisfaction with vision, as well as questions assessing performance in specific daily activities. Each question has multiple predefined response categories ranging from "very great difficulty" to "no difficulty". One question has response categories ranging from "very dissatisfied" to "very satisfied". All questions have a "can't say"-response category. Each response will be translated to a numerical value used to score the participants.

In addition to the Catquest-7SF, the questionnaire used will also include questions related to satisfaction with the surgical approach (same day or delayed) and experiences with and knowledge of complex visual hallucinations.

The additional questions about complex visual hallucinations are used to measure prevalence and knowledge of Charles Bonnet Syndrome among participants referred to elective cataract surgery.

The study is a prospective, randomized cohort study and will include 300 consecutive patients referred to our department for elective bilateral cataract surgery. Eligible patients who provide consent will be randomly allocated in a group of either same day bilateral surgery or surgery on two days separated by one week. In case of serious surgical complications in the same day group, surgery of the second eye will be postponed and the participant will be placed in a new, separate group.

During a preoperative visit to the department, participants will fill out the questionnaire regarding vision and be subjected to the routine clinical ophthalmic examination which includes biometry and refraction status. One day post-surgery, participants will be contacted by phone regarding their vision. One-week post-surgery, participants will undergo a check-up visit that includes the same examinations as the preoperative visit, except for biometry. Three months post-surgery, participants will once again be contacted by phone or letter and asked to fill out the questionnaire again.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for bilateral cataract surgery with monofocal intraocular lens implantation in the bag.
* Patients who agree to be randomly allocated to either ISBCS or DSBCS

Exclusion Criteria:

* Patients at risk of intra- og postoperative complications or where delayed visual rehabilitation is expected (e.g. glaucoma, anterior chamber depth 2,3 or less, corneal endothelial dystrophy)
* Patients with axial lengths < 21 mm or > 27 mm
* Patients in need of immediate surgery
* Patients only eligible to one group, e.g. those requiring general anesthesia where ISBCS is the preferred approach
* Patients unable to read, understand or fill out the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in patient reported visual function outcome following either ISBCS or DSBCS | Baseline at the preoperative visit, 1 week post-surgery, and 3 months post-surgery
  Change in participant satisfaction in regards to visual function measured using the Catquest 7-SF questionnaire at the preoperative visit as well as 1 week and 3 months after either ISBCS or 2nd eye surgery in DSBCS

SECONDARY OUTCOMES:
Objective change in visual acuity | At the preoperative visit and 1 week after ISBCS or 2nd eye surgery in DSBCS
  Measured using autorefractor
Objective change in refraction status | At the preoperative visit and 1 week after ISBCS or 2nd eye surgery in DSBCS
  Measured using autorefractor
Intraocular pressure (IOP) | At the preoperative visit and 1 week after ISBCS or 2nd eye surgery in DSBCS
  Measured using I-Care Tonometry
Complications | Intraoperatively, one day after surgery and up to one week after ISBCS or 2nd eye surgery in DSBCS
  Incidence of intraoperative and postoperative complications
Presence of corneal edema | One week after ISBCS or 2nd eye surgery in DSBCS
  Determined during clinical examination using slit lamp
Presence of Charles Bonnet Syndrome | At the preoperative visit
  Participants will be asked if they have experienced complex, visual hallucinations during the time in which their vision has been affected by cataract. In case of presence of complex visual hallucinations, patients will be further interviewed regarding the characteristics of the hallucinations.
Knowledge of Charles Bonnet Syndrome | At the preoperative visit
  Participants will be asked about previous knowledge of hallucinations caused by loss of vision.

CONTACTS AND LOCATIONS:
Overall Officials: Amardeep Singh, MD, PhD, Study Director — Dpt. of Ophthalmology, Rigshospitalet-Glostrup; University of Copenhagen; Mads Assenholt Nielsen, Principal Investigator — Dpt. of Ophthalmology, Rigshospitalet-Glostrup; University of Copenhagen
Locations (1):
- Department of Ophthalmology, Rigshospitalet-Glostrup, Glostrup Municipality, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arshinoff SA, Odorcic S. Same-day sequential cataract surgery. Curr Opin Ophthalmol. 2009 Jan;20(1):3-12. doi: 10.1097/ICU.0b013e32831b6daf. PMID 19077823
- [Background] Arshinoff SA. Same-day cataract surgery should be the standard of care for patients with bilateral visually significant cataract. Surv Ophthalmol. 2012 Nov;57(6):574-9. doi: 10.1016/j.survophthal.2012.05.002. Epub 2012 Sep 18. PMID 22995967
- [Background] Arshinoff SA, Claoue C, Mehta C, Johanssen B, Mota SH. Bilateral Pseudomonas endophthalmitis after immediately sequential bilateral cataract surgery: primum non nocere. Arq Bras Oftalmol. 2020 Aug;83(4):346-349. doi: 10.5935/0004-2749.20200073. Epub 2020 Jul 29. No abstract available. PMID 32756782
- [Background] Cetinkaya S, Dadaci Z, Aksoy H, Acir NO, Yener HI, Kadioglu E. Toxic anterior-segment syndrome (TASS). Clin Ophthalmol. 2014 Oct 9;8:2065-9. doi: 10.2147/OPTH.S71541. eCollection 2014. PMID 25336907
- [Background] Coyle D, Drummond M. The economic burden of glaucoma in the UK. The need for a far-sighted policy. Pharmacoeconomics. 1995 Jun;7(6):484-9. doi: 10.2165/00019053-199507060-00003. No abstract available. PMID 10155334
- [Background] Hartney KE, Catalano G, Catalano MC. Charles Bonnet syndrome: are medications necessary? J Psychiatr Pract. 2011 Mar;17(2):137-41. doi: 10.1097/01.pra.0000396067.87343.fb. PMID 21430494
- [Background] Henderson BA, Schneider J. Same-day cataract surgery should not be the standard of care for patients with bilateral visually significant cataract. Surv Ophthalmol. 2012 Nov;57(6):580-3. doi: 10.1016/j.survophthal.2012.05.001. Epub 2012 Sep 18. PMID 22995968
- [Background] Herrinton LJ, Liu L, Alexeeff S, Carolan J, Shorstein NH. Immediate Sequential vs. Delayed Sequential Bilateral Cataract Surgery: Retrospective Comparison of Postoperative Visual Outcomes. Ophthalmology. 2017 Aug;124(8):1126-1135. doi: 10.1016/j.ophtha.2017.03.034. Epub 2017 Apr 21. PMID 28438415
- [Background] Jones L, Ditzel-Finn L, Potts J, Moosajee M. Exacerbation of visual hallucinations in Charles Bonnet syndrome due to the social implications of COVID-19. BMJ Open Ophthalmol. 2021 Feb 11;6(1):e000670. doi: 10.1136/bmjophth-2020-000670. eCollection 2021. PMID 33628948
- [Background] Leivo T, Sarikkola AU, Uusitalo RJ, Hellstedt T, Ess SL, Kivela T. Simultaneous bilateral cataract surgery: economic analysis; Helsinki Simultaneous Bilateral Cataract Surgery Study Report 2. J Cataract Refract Surg. 2011 Jun;37(6):1003-8. doi: 10.1016/j.jcrs.2010.12.050. PMID 21596243
- [Background] Lundstrom M, Albrecht S, Roos P. Immediate versus delayed sequential bilateral cataract surgery: an analysis of costs and patient value. Acta Ophthalmol. 2009 Feb;87(1):33-8. doi: 10.1111/j.1755-3768.2008.01343.x. Epub 2008 Sep 11. PMID 18786128
- [Background] Lundstrom M, Pesudovs K. Catquest-9SF patient outcomes questionnaire: nine-item short-form Rasch-scaled revision of the Catquest questionnaire. J Cataract Refract Surg. 2009 Mar;35(3):504-13. doi: 10.1016/j.jcrs.2008.11.038. PMID 19251145
- [Background] Morley AM, Murdoch I. The future of glaucoma clinics. Br J Ophthalmol. 2006 May;90(5):640-5. doi: 10.1136/bjo.2005.085522. PMID 16622096
- [Background] Niazi S, Krogh Nielsen M, Singh A, Sorensen TL, Subhi Y. Prevalence of Charles Bonnet syndrome in patients with age-related macular degeneration: systematic review and meta-analysis. Acta Ophthalmol. 2020 Mar;98(2):121-131. doi: 10.1111/aos.14287. Epub 2019 Oct 26. PMID 31654492
- [Background] Nielsen E, Lundstrom M, Pesudovs K, Hjortdal J. Validation of Catquest-9SF in Danish: developing a revised form of the Catquest-9SF - the Danish Catquest-7SF. Acta Ophthalmol. 2019 Mar;97(2):173-177. doi: 10.1111/aos.13921. Epub 2018 Sep 21. PMID 30242976
- [Background] Singh R, Dohlman TH, Sun G. Immediately sequential bilateral cataract surgery: advantages and disadvantages. Curr Opin Ophthalmol. 2017 Jan;28(1):81-86. doi: 10.1097/ICU.0000000000000327. PMID 27684294
- [Background] Singh A, Sorensen TL. The prevalence and clinical characteristics of Charles Bonnet Syndrome in Danish patients with neovascular age-related macular degeneration. Acta Ophthalmol. 2012 Aug;90(5):476-80. doi: 10.1111/j.1755-3768.2010.02051.x. Epub 2010 Nov 25. PMID 21106047
- [Background] Singh A, Sorensen TL. Charles Bonnet syndrome improves when treatment is effective in age-related macular degeneration. Br J Ophthalmol. 2011 Feb;95(2):291-2. doi: 10.1136/bjo.2010.179465. Epub 2010 Aug 23. No abstract available. PMID 20733019
- [Background] Smith CS, Nichols J, Riaz KM. Remission of Charles Bonnet syndrome after cataract extraction. Can J Ophthalmol. 2018 Dec;53(6):e221-e222. doi: 10.1016/j.jcjo.2018.01.036. Epub 2018 Apr 2. No abstract available. PMID 30502996
- [Background] Subhi Y, Schmidt DC, Bach-Holm D, Kolko M, Singh A. Prevalence of Charles Bonnet syndrome in patients with glaucoma: a systematic review with meta-analyses. Acta Ophthalmol. 2021 Mar;99(2):128-133. doi: 10.1111/aos.14567. Epub 2020 Aug 4. PMID 32749787
- [Background] Tatham A, Brookes JL. 'Bilateral same-day cataract surgery should routinely be offered to patients' - no. Eye (Lond). 2012 Aug;26(8):1033-5. doi: 10.1038/eye.2012.92. Epub 2012 May 25. No abstract available. PMID 22627481
- [Background] Denniston AK, Holland GN, Kidess A, Nussenblatt RB, Okada AA, Rosenbaum JT, Dick AD. Heterogeneity of primary outcome measures used in clinical trials of treatments for intermediate, posterior, and panuveitis. Orphanet J Rare Dis. 2015 Aug 19;10:97. doi: 10.1186/s13023-015-0318-6. PMID 26286265
- [Background] European Glaucoma Society: Terminology and guidelines for glaucoma, 3rd edn (2008). Savona, Italy: Editrice Dogma S.r.l.
- [Background] Kessel L, Andresen J, Erngaard D, Flesner P, Tendal B, Hjortdal J. Immediate Sequential Bilateral Cataract Surgery: A Systematic Review and Meta-Analysis. J Ophthalmol. 2015;2015:912481. doi: 10.1155/2015/912481. Epub 2015 Aug 17. PMID 26351576
- [Background] Lundstrom M, Fregell G, Sjoblom A. Vision related daily life problems in patients waiting for a cataract extraction. Br J Ophthalmol. 1994 Aug;78(8):608-11. doi: 10.1136/bjo.78.8.608. PMID 7918286
- [Background] Tuulonen A & Sintonen H. Health economics, cost-effectiveness and glaucoma care. Grehn F & Stamper R (eds) Glaucoma 2006. Berlin: Springer, 123-133